CLINICAL TRIAL: NCT01665313
Title: Comparison of Performance, Attention, and Emotion of Physician Before and After Outpatient Clinic Session
Brief Title: Comparison of Attention of Physician After Outpatient Clinic
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: attention_SNUH
Record Dates: First submitted 2012-07-08; First posted 2012-08-15 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Disturbance of Activity and Attention
Keywords: attention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- participants: Full-time faculty with morning and afternoon outpatient clinics on the same day in SNUH

SUMMARY:
The attention and clinical performance of physician might be decreased after outpatient clinic session compared to those measured before outpatient clinic.

DETAILED DESCRIPTION:
A large body of data shows that fatigue impairs human performance. Additionally, many studies have provided evidence that fatigue can worsen mood, as indicated by increased scores on measures of depression, anxiety, confusion, and anger. In this context, we examined attentional and emotional changes in physicians after they completed an overwhelming outpatient clinic in a university-affiliated tertiary referral hospital in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* physicians with outpatient clinic sessions in Seoul National University Hospital
* age 30~59
* internal part or external part

Exclusion Criteria:

* physicians who do not agree to participate in the study
* physicians who are taking drugs known to affect the sleep/wake cycle or daytime alertness
* physicians who have current psychiatric illness or sleep disorder

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: physicians with outpatient clinic sessions in Seoul National University Hospital
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
difference of response time in PVT(Psychomotor vigilance task) before and after outpatient clinic session | change from baseline in response time in PVT after opd session (average 7hours)

SECONDARY OUTCOMES:
frequency of physician's clinical mistakes during morning and afternoon session in outpatient clinic | for the duration of opd session, average up to 7hours

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Joon Yim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea